CLINICAL TRIAL: NCT04911270
Title: A Pharmacokinetic Study to Evaluate the Use of a Novel Clinical Decision Support Tool, Lyv, in Achieving AUC24/MIC > 400 in Pediatric Patients on Vancomycin
Brief Title: Clinical Decision Support Tool for Vancomycin Dosing in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Center for Translational Medicine at the School of Pharmacy (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Siddhartha Dante, Assistant Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00093185; T32HD087969 (NIH)
Record Dates: First submitted 2021-05-24; First posted 2021-06-03 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Gram-Positive Bacterial Infections; Vancomycin; Pharmacokinetics; Pharmacodynamics
Keywords: computer decision support; gram positive bacterial infections; sepsis; vancomycin
MeSH Terms: conditions — Gram-Positive Bacterial Infections; Sepsis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The intervention group includes pediatric patients that will be started on intravenous (IV) vancomycin. Once consent is obtained, their age, weight, length, sex, serum creatinine will be entered into Lyv which will generate a dose for the patient. Levels will be drawn intermittently and dosage will be adjusted accordingly. This interventional group will be compared to matched historical controls who were treated with IV vancomycin with dosage adjustments based on trough levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group- Computer Decision Support Tool (Experimental): Patients enrolled in the study will be started on IV vancomycin which will be dosed based on the LYV CDS tool, which will dose patients based on AUC24/MIC. Dosing will be adjusted based on vancomycin levels that will be drawn throughout the hospital stay.
  All patients prospectively enrolled into this study will be in the intervention group. Results will be compared to the retrospectively matched historical controls.
  Interventions: Device: Computer Decision Support Tool Intervention Group
- Matched Historical Controls (Other): Match historical controls are patients that were on IV vancomycin with dose adjustments based on vancomycin trough levels. Patients in this study arm will be retrospective patients that will be matched with the intervention group.
  Interventions: Other: Matched Historical Controls

INTERVENTIONS:
Device: Computer Decision Support Tool Intervention Group — Computer Decision Support Tool using Bayesian estimation to dose IV vancomycin in pediatric patients using AUC24/MIC
  Other Names: Lyv
  Arms: Intervention Group- Computer Decision Support Tool
Other: Matched Historical Controls — Vancomycin dosing based on standard hospital methods, with dose adjustments based on vancomycin trough targets
  Other Names: standard of care
  Arms: Matched Historical Controls

SUMMARY:
This study will evaluate the pharmacokinetic and pharmacodynamic dosing properties of intravenous vancomycin in pediatric patients using a novel computer decision support (CDS) tool called Lyv. Dosing will be individualized based on AUC24/MIC. The results will be compared to matched historical controls.

DETAILED DESCRIPTION:
This study is a prospective pharmacokinetic study of pediatric patients receiving IV vancomycin at the University of Maryland. Patients may be in the Pediatric Intensive Care Unit (PICU), Neonatal Intensive Care Unit (NICU), the Intermediate Care Unit (IMC) or the general pediatric ward.

The study design will be comparing historical controls, who are retrospective patients that had IV vancomycin dosed based on pharmacists' calculations, to prospective patients who will have vancomycin dosing based on a clinical decision support tool.

Patients requiring IV vancomycin therapy will be selected on the basis of inclusion and exclusion criteria. The study procedures will be explained to all patients and written informed consent will be obtained from each subject prior to enrollment.

Historical controls will be selected based on the same inclusion and exclusion criteria to minimize bias. Full HIPPA waiver will be used for these patients.

All patients who consent to enrolling in the study will have vancomycin dosing based on the Clinical Decision Support (CDS) tool. Results will be compared to historical controls. Patients must be enrolled within the first 24 hours of initiation of vancomycin.

Conventional hospital method- Historical Controls (standard of care)- retrospective:

Data will be collected from patients who were initiated on vancomycin using doses determined by the population parameter calculations. These patients will have a minimum of one serum creatinine documented. Trough concentrations of vancomycin will typically be collected 30 minutes prior to the 3rd dose. Multiple troughs may be collected and will be used for analysis.

Clinical Decision Support method (intervention group)- prospective:

Patient information will be entered into the decision support system to calculate vancomycin dose to be initiated in patients after consent is obtained. After enrollment into the study, the patients serum creatinine level, age (post-menstrual age if less than one year of age), sex, weight in kilograms, and height in centimeters will be entered into the CDS tool and a suggested dose (in mg/kg) and dosing interval (in hours) will be recommended. All doses recommended by the CDS tool must be approved by the pharmacist. If the dosing recommendation was, for any reason, overridden, then it will be recorded in the case report forms. The pharmacist will also calculate the AUC24/MIC manually. The proposed dose by the CDS tool should be within a 20% margin of error of the manually calculated dose. The pharmacist will have the option of using the proposed dosing regimen or standard dosing if there is concern with the proposed dose.

Once vancomycin has been infused, there will be one to two random levels drawn within the first 24 hours, and most optimally at least one level drawn prior to the second dose. Timing of these blood draws can vary and can be paired with other blood draws that are occurring at the same time. This information will then be entered into the CDS tool and the following dose(s) will be calculated. Standard trough levels will also be drawn at the discretion of the clinician and will also be used as data points in the CDS tool.

These levels will be entered back into the decision support system to determine if the target AUC/MIC is/will be attained and if necessary, calculate the new dose. If a new dose was required, another level will again be taken after the newly calculated dose was administered.

Subjects will participate in the study for up to 7 days. For all subjects, the number of blood samples collected for research-related vancomycin level determination will not exceed 5.

Serum Samples:

Blood samples will be obtained by nursing or medical staff or whoever routinely collects blood samples as part of the standard of care in that unit. When possible, blood samples obtained as part of routine clinical care for other laboratory assessments will be used in order to minimize the risk to the subjects. Samples can be drawn from a peripherally inserted central catheter (PICC), peripheral IV, central line, arterial line, or a separate blood draw. If it is drawn from the same line that was infusing the vancomycin, adequate blood waste must occur. This includes 3 mL if <2 years old, or 5 mL if >2 years old. Serum samples will be sent to the University of Maryland laboratory. Serum vancomycin levels can only be reported by the laboratory if >5 mg/L. If it is less than 5 it will be entered as 0 into the CDS.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized infants and children from postmenstrual age of 38 weeks to age 19 years Requiring IV vancomycin, regardless of indication
* Parent or legally authorized representative is willing to provide permission and sign the informed consent document; subjects assent, when appropriate
* Hospitalized neonates, infants, children, adolescents who require, but have not been initiated on intravenous vancomycin therapy

Exclusion Criteria:

* Patients who had received vancomycin during previous 2 weeks
* Patients with end-stage renal disease, receiving hemodialysis or receiving continuous renal replacement therapy
* On oral or intraperitoneal vancomycin
* Receiving extracorporeal therapy, including extracorporeal membrane oxygenation, continuous renal replacement therapy, and extracorporeal liver support
* Will only receive a single dose of vancomycin
* Known to be pregnant
* Is brain dead or has suspected brain death

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
AUC24/MIC target attainment of vancomycin after first dose using the clinical decision support tool compared to dosing using the current hospital method | 2-6 hours post first dose
  Vancomycin level will be drawn after first dose of antibiotic. The level will be entered into the CDS tool and AUC24/MIC target attainment will be generated. If the level is not in range, the CDS tool will generate a new dose for future doses.

SECONDARY OUTCOMES:
To characterize vancomycin pharmacokinetics and evaluate the factors that affect variability in achievement of an AUC24/MIC > 400 in pediatric patients | From start to end of antibiotic therapy, or a max of 7 days
  Factors such as weight, height, serum creatinine, fluid status, vancomycin dose, and vancomycin level will be documented. These factors will be compared to those in the historical controls.
To evaluate the incidence of nephrotoxicity for dosing vancomycin using the decision support tool compared to dosing using the current hospital method | From start to end of antibiotic therapy, or a max of 7 days
  Evaluate creatinine levels prior to starting, during, and after vancomycin therapy. Will also document concomitant medications, fluid balance, and illness and compare to historical controls.
  Using creatinine levels, will assess AKI by KDIGO AKI definition.
To evaluate the accuracy of the clinical decision support system in predicting the AUC24/MIC | From start to end of antibiotic therapy, or a max of 7 days
  Vancomycin levels will be drawn at random times throughout antibiotic therapy and will be entered into CDS tool and target attainment will be generated. These measurements will be documented, as well as a percentage from target, if target is not obtained

OTHER OUTCOMES:
The number of dose changes before getting to the therapeutic dose, defined as the dose achieving AUC24/MIC > 400 | From start to end of antibiotic therapy, or a max of 7 days
  Each vancomycin dose, vancomycin level, number of dose changes, and percent difference from goal AUC24/MIC will be documented and assessed. Dose changes will be compared to historical controls.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu C, Bayer A, Cosgrove SE, Daum RS, Fridkin SK, Gorwitz RJ, Kaplan SL, Karchmer AW, Levine DP, Murray BE, J Rybak M, Talan DA, Chambers HF. Clinical practice guidelines by the infectious diseases society of america for the treatment of methicillin-resistant Staphylococcus aureus infections in adults and children: executive summary. Clin Infect Dis. 2011 Feb 1;52(3):285-92. doi: 10.1093/cid/cir034. PMID 21217178
- [Background] Iwamoto M, Mu Y, Lynfield R, Bulens SN, Nadle J, Aragon D, Petit S, Ray SM, Harrison LH, Dumyati G, Townes JM, Schaffner W, Gorwitz RJ, Lessa FC. Trends in invasive methicillin-resistant Staphylococcus aureus infections. Pediatrics. 2013 Oct;132(4):e817-24. doi: 10.1542/peds.2013-1112. Epub 2013 Sep 23. PMID 24062373
- [Background] Gerber JS, Coffin SE, Smathers SA, Zaoutis TE. Trends in the incidence of methicillin-resistant Staphylococcus aureus infection in children's hospitals in the United States. Clin Infect Dis. 2009 Jul 1;49(1):65-71. doi: 10.1086/599348. PMID 19463065
- [Background] Moise-Broder PA, Forrest A, Birmingham MC, Schentag JJ. Pharmacodynamics of vancomycin and other antimicrobials in patients with Staphylococcus aureus lower respiratory tract infections. Clin Pharmacokinet. 2004;43(13):925-42. doi: 10.2165/00003088-200443130-00005. PMID 15509186
- [Background] Giachetto GA, Telechea HM, Speranza N, Oyarzun M, Nanni L, Menchaca A. Vancomycin pharmacokinetic-pharmacodynamic parameters to optimize dosage administration in critically ill children. Pediatr Crit Care Med. 2011 Nov;12(6):e250-4. doi: 10.1097/PCC.0b013e3181fe4047. PMID 21057350
- [Background] Gous AG, Dance MD, Lipman J, Luyt DK, Mathivha R, Scribante J. Changes in vancomycin pharmacokinetics in critically ill infants. Anaesth Intensive Care. 1995 Dec;23(6):678-82. doi: 10.1177/0310057X9502300603. PMID 8669599
- [Background] Le J, Bradley JS, Murray W, Romanowski GL, Tran TT, Nguyen N, Cho S, Natale S, Bui I, Tran TM, Capparelli EV. Improved vancomycin dosing in children using area under the curve exposure. Pediatr Infect Dis J. 2013 Apr;32(4):e155-63. doi: 10.1097/INF.0b013e318286378e. PMID 23340565
- [Background] Kaddourah A, Basu RK, Bagshaw SM, Goldstein SL; AWARE Investigators. Epidemiology of Acute Kidney Injury in Critically Ill Children and Young Adults. N Engl J Med. 2017 Jan 5;376(1):11-20. doi: 10.1056/NEJMoa1611391. Epub 2016 Nov 18. PMID 27959707
- [Background] Heil EL, Claeys KC, Mynatt RP, Hopkins TL, Brade K, Watt I, Rybak MJ, Pogue JM. Making the change to area under the curve-based vancomycin dosing. Am J Health Syst Pharm. 2018 Dec 15;75(24):1986-1995. doi: 10.2146/ajhp180034. Epub 2018 Oct 17. No abstract available. PMID 30333114
- [Background] Hughes DM, Goswami S, Keizer RJ, Hughes MA, Faldasz JD. Bayesian clinical decision support-guided versus clinician-guided vancomycin dosing in attainment of targeted pharmacokinetic parameters in a paediatric population. J Antimicrob Chemother. 2020 Feb 1;75(2):434-437. doi: 10.1093/jac/dkz444. PMID 31670812